CLINICAL TRIAL: NCT01570075
Title: Radiofrequency Ablation Versus Liver Resection for Elderly Patients With Hepatocellular Carcinoma (HCC) Within the Milan Criteria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, professor, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HCC17
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; RFA; HR
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA group (Experimental): For RFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Interventions: Procedure: HR
- HR group (Experimental): SR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: HR — SR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure.
  Other Names: hepatic resection; surgical resection
  Arms: RFA group
Procedure: RFA — For PRFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Other Names: percutaneous ablation
  Arms: HR group

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cancer, and it is the third commonest global cause of cancer-related death. With an increase in life-expectancy of the general population, the number of elderly with HCC is expected to increase. Current curative treatment options for HCC include: liver transplantation, liver resection (LR) and local ablation therapy. Liver transplantation is a good treatment for HCC within the Milan criteria (single HCC ≤ 5 cm or up to 3 nodules each < 3 cm). As a consequence of the lack of liver donors, one relative contraindication for liver transplantation is age over 65 years, or the protocol requires elderly patients to have very good general health before they can be put on a transplant list. Transcatheter arterial chemoembolization (TACE) is used more commonly for the treatment of intermediate and advanced-staged HCC, while liver resection and local ablation therapy are used for early-staged HCC. Amongst the local ablative therapies, radiofrequency ablation (RFA) is most widely used. It has the advantage of minimally invasiveness, making it the first-line treatment for small HCC in patients with compromised liver function or associated severe medical conditions.

Elderly patients are more likely to have poor general conditions and associated medical diseases. RFA has the advantage of being less invasive and it causes less pain, less blood loss and earlier recovery than LR. On the other hand, incomplete ablation of HCC and tumor track seeding may happen. Several studies have demonstrated the safety of LR for elderly patients. There is no good evidence in the medical literature to support whether RFA or LR is a better treatment for elderly patients with HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common cancer, and it is the third commonest global cause of cancer-related death. With an increase in life-expectancy of the general population, the number of elderly with HCC is expected to increase. Current curative treatment options for HCC include: liver transplantation, liver resection (LR) and local ablation therapy. Liver transplantation is a good treatment for HCC within the Milan criteria (single HCC ≤ 5 cm or up to 3 nodules each < 3 cm). As a consequence of the lack of liver donors, one relative contraindication for liver transplantation is age over 65 years, or the protocol requires elderly patients to have very good general health before they can be put on a transplant list. Transcatheter arterial chemoembolization (TACE) is used more commonly for the treatment of intermediate and advanced-staged HCC, while liver resection and local ablation therapy are used for early-staged HCC. Amongst the local ablative therapies, radiofrequency ablation (RFA) is most widely used. It has the advantage of minimally invasiveness, making it the first-line treatment for small HCC in patients with compromised liver function or associated severe medical conditions.

Elderly patients are more likely to have poor general conditions and associated medical diseases. RFA has the advantage of being less invasive and it causes less pain, less blood loss and earlier recovery than LR. On the other hand, incomplete ablation of HCC and tumor track seeding may happen. Several studies have demonstrated the safety of LR for elderly patients. There is no good evidence in the medical literature to support whether RFA or LR is a better treatment for elderly patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 - 85 years;
2. HCC within the Milan criteria (single HCC ≤ 5 cm or up to 3 nodules each ≤3 cm);
3. resectable disease, which is defined as the possibility of completely removing all tumors and retaining a sufficient liver remnant to maintain liver function, as assessed by our surgery team;
4. Eastern Co-operative Oncology Group performance (ECOG) status 0 ;

Exclusion Criteria:

1. severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
2. the presence of vascular invasion or extrahepatic spread on imaging;
3. Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding, or hepatic encephalopathy;
4. previous treatment.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
disease-free survival | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-set University, Guangzhou, Guangdong, China